CLINICAL TRIAL: NCT00354198
Title: Clinical Efficacy of Combined Pentoxifylline and Conventional Immunosuppressive Regimens on Patients With Rapidly Progressive Glomerulonephritis
Brief Title: Efficacy of Pentoxifylline on Rapidly Progressive Glomerulonephritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: short of participants
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 941008
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-10

CONDITIONS: Glomerulonephritis
Keywords: rapidly progressive glomerulonephritis; pentoxifylline
MeSH Terms: conditions — Glomerulonephritis | interventions — Pentoxifylline; Adrenal Cortex Hormones; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- corticosteroids (Active Comparator): [intravenous pulse methylprednisolone (15 mg/kg/day or a maximum of 1 g/day) x 3 days + oral prednisolone (0.5-1.0 mg/kg/day) for 27 days] x 3 courses
  Interventions: Drug: corticosteroids
- pentoxifylline + corticosteroids (Experimental): [intravenous pulse methylprednisolone (15 mg/kg/day or a maximum of 1 g/day) x 3 days + oral prednisolone (0.5-1.0 mg/kg/day) for 27 days] x 3 courses + intravenous infusion of pentoxifylline (0.33-0.66 mg/kg/h) x 7 days + oral pentoxifylline (400-800 mg/day) from days 8 to 90
  Interventions: Drug: pentoxifylline; Drug: corticosteroids

INTERVENTIONS:
Drug: pentoxifylline — intravenous pentoxifylline (0.33-0.66 mg/kg/h from days 1 to 7) followed by oral pentoxifylline 400-800 mg/day (from days 8-90). The dose of intravenous pentoxifylline will be determined by estimated GFR, patients whose GFRs are 30-59 ml/min/1.73 m2 will be given 0.66 mg/kg/h, and those below 30 ml/min/1.73 m2 will be given 0.33 mg/kg/h. The oral dose of pentoxifylline will also be determined by estimated GFR. Patients whose estimated GFRs are between 30-59 ml/min/1.73 m2 will be given 800 mg/day, and those below 30 ml/min/1.73 m2 will be given 400 mg/day.
  Other Names: Trental
  Arms: pentoxifylline + corticosteroids
Drug: corticosteroids — intravenous methylprednisolone (15 mg/kg/day or a maximum of 1 g/day) x 3 days + oral prednisolone (0.5-1.0 mg/kg/day) for 27 days] x 3 courses
  Other Names: Solu-medrol, Predonin

SUMMARY:
We have recently demonstrated that pentoxifylline (PTX) has the potential to treat severe glomerular inflammation in a rat model of accelerated anti-glomerular basement membrane (GBM) glomerulonephritis. This study aims to investigate the therapeutic effects of combined PTX and conventional immunosuppressive regimens on patients with rapidly progressive glomerulonephritis.

DETAILED DESCRIPTION:
Corticosteroids and cytotoxic agents such as cyclophosphamide remain the most commonly used regimens for crescentic glomerulonephritis. However, their use is often limited by adverse effects, most notably life-threatening opportunistic infections due to generalized immunosuppression. Over the past decade, a number of novel experimental therapeutic agents have been shown to ameliorate the severity of experimental crescentic glomerulonephritis. Unfortunately, none of these measures is currently available for clinical use. Other potential agents such as mycophenolate, cyclosporin, and tacrolimus , while clinically available, share similar adverse effects with corticosteroid- and cyclophosphamide-based regimens. PTX is a methylxanthine phosphodiesterase inhibitor that has been widely used to treat peripheral vascular diseases and cerebrovascular disorders. In addition to its well-known hemorheologic activity, accumulating evidence suggests that PTX also possesses potent anti-inflammatory and/or immunoregulatory activities. For examples, PTX has shown its efficacy in different animal models of renal diseases where tumor necrosis factor (TNF)-alpha, monocyte chemoattractant protein (MCP)-1, or intercellular adhesion molecule-1 is involved. Moreover, clinical trials in patients with diabetic nephropathy and membranous glomerulonephritis have shown that PTX can lower endogenous TNF-alpha and attenuate proteinuria. These data raise the possibility that PTX may have promise as an anti-inflammatory agent via its ability to antagonize inflammatory mediators. Consistent with this idea, we have demonstrated this potential usefulness of PTX in a rat model of accelerated anti-GBM glomerulonephritis. More recently, we have reported that PTX is capable of inhibiting proteinuria via renal MCP-1 production in subnephrotic primary glomerular diseases. In this study, we aim to investigate the potential benefit of combined PTX and conventional immunosuppressive regimens, compared to conventional immunosuppressive therapy, in patients with rapidly progressive glomerulonephritis.

This study is a randomized, open-label, comparative study. Group A is treated by three monthly standard intravenous pulse-dose methylprednisolone (15 mg/kg/day or a maximum of 1 g/day from days 1 to 3) followed by oral prednisolone 0.5-1.0 mg/kg/day (from days 4-30). Group B is treated by the same corticosteroid regimen plus intravenous PTX (0.33-0.66 mg/kg/h from days 1 to 7) followed by oral PTX 400-800 mg/day (from days 8-90). The dose of intravenous PTX will be determined by estimated GFR, patients whose GFRs are 30-59 ml/min/1.73 m2 will be given 0.66 mg/kg/h, and those below 30 ml/min/1.73 m2 will be given 0.33 mg/kg/h. The oral dose of PTX will also be determined by estimated GFR. Patients whose estimated glomerular filtration rates (GFRs) are between 30-59 ml/min/1.73 m2 will be given 800 mg/day, and those below 30 ml/min/1.73 m2 will be given 400 mg/day. If the patients cannot tolerate oral medications, either PTX or corticosteroids can be administered intravenously until patients can resume oral intakes. Serum and single-voided urine specimens will be collected at the hospital before initiation of therapy (day 0), and at days 8, 15, 30, and 90 after the commencement of therapy. Renal function will be calculated by Cockcroft-Gault and simplified Modification of Diet in Renal Disease formula. All biochemical and immunological analyses will be performed by the Department of Laboratory Medicine, National Taiwan University Hospital. Serum and urine samples will be measured for inflammatory mediators using commercial ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* biopsied-proved crescentic glomerulonephritis, with rapidly progressive renal failure

Exclusion Criteria:

* Anti-GBM disease, Dialysis-dependency or pulmonary hemorrhage, History of allergy to pentoxifylline, Females are nursing or pregnant, Congestive heart failure, Unstable angina, myocardial infarction, coronary artery bypass graft surgery, percutaneous coronary intervention, within the past 6 months prior to signing the informed consent form, Cerebral hemorrhage within the past 6 months prior to signing the informed consent form, Retinal hemorrhage within the past 6 months prior to signing the informed consent form, Known or suspected secondary hypertension, Uncontrolled hypertension or diabetes, Liver cirrhosis or hepatic dysfunction as defined by liver enzymes > 2 times the upper limit of the normal range, Biliary obstructive disorders, Active malignancy or infection

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-08; Primary Completion 2009-08 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
initiation of acute dialysis or doubling of serum creatinine levels | 3 months

SECONDARY OUTCOMES:
end-stage renal disease (ESRD) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Ming Chen, M.D., Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan